MEDICAL RECORD

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

Adult Patient or

· Parent, for Minor Patient

INSTITUTE:

National Cancer Institute

STUDY NUMBER:

11-C-0016

PRINCIPAL INVESTIGATOR:

Daniel H. Fowler, M.D.

STUDY TITLE:

Rapamycin-Resistant T Cell Therapy of Multiple Myeloma: Relapse Prevention and

Relapse Therapy

Continuing Review Approved by the IRB on 12/19/16

Amendment Approved by the IRB on 02/16/17 (O)

Date posted to web: 03/03/17

Addendum to 11-C-0016

This addendum provides new information about the study "Rapamycin-Resistant T Cell Therapy of Multiple Myeloma: Relapse Prevention and Relapse Therapy" on which you are enrolled. The information in the consent you signed previously is unchanged.

The NIH Clinical Center Pharmaceutical Development Service (PDS) helps prepare the stem cells used in this study. The PDS was recently closed down by NIH leadership after a vial of contaminated material was discovered on another study just before it was supposed to be given to a research participant. The PDS is undergoing a full review and changes are being made to make sure that processes are in place to prevent anything like this from happening again. The FDA and NIH decided that it might be better and safer to make an exception to the PDS shutdown for some research studies as long as those decisions are made on a case by case basis. The stem cells used for T cell transplant received one of those exceptions because it would be potentially very harmful for you to not receive the cells. Before giving the exception, the FDA and NIH determined that the risk to you from receiving the stem cells that includes the portions made by the PDS, before all of the reviews and changes to the PDS are finished, is extremely low.

 Adult Patient or NIH-2514-1 (07-09) · Parent, for Minor Patient

P.A.: 09-25-0099

File in Section 4: Protocol Consent (2)

MEDICAL RECORD

## CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

· Adult Patient or

Parent, for Minor Patient

STUDY NUMBER: 11-C-0016

CONTINUATION: page 2 of 2 pages

| COMPLETE APPROPRIATE ITEM(S) BELOW: | |
|---|---|
| A. Adult Patient's Consent | B. Parent's Permission for Minor Patient. |
| I have read the explanation about this study | I have read the explanation about this study |
| and have been given the opportunity to discuss | and have been given the opportunity to discuss |
| it and to ask questions. I hereby consent to | it and to ask questions. I hereby give |
| take part in this study. | permission for my child to take part in this |
| | study. |
| | (Attach NIH 2514-2, Minor's Assent, if applicable.) |
| Signature of Adult Patient/ Date | Signature of Deposit/5)/ Cyandian Deta |
| Legal Representative | Signature of Parent(s)/ Guardian Date |
| , | |
| Print Name | Print Name |
| C. Child's Verbal Assent (If Applicable) The information in the above consent was described to my child and my child agrees to participate in the study. | |
| Signature of Parent(s)/Guardian Date | Print Name |
| THIS CONSENT DOCUMENT HAS BEEN APPROVED FOR USE FROM DECEMBER 19, 2016 THROUGH DECEMBER 18, 2017. | |
| Signature of Investigator Date | Signature of Witness |
| Date Date | Signature of Witness Date |
| Print Name | Print Name |

PATIENT IDENTIFICATION

CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY (Continuation Sheet)

Adult Patient or

· Parent, for Minor Patient

NIH-2514-1 (07-09) P.A.: 09-25-0099

File in Section 4: Protocol Consent